CLINICAL TRIAL: NCT04498832
Title: Immunogenicity and Safety of High-Dose Quadrivalent Influenza Vaccine (SP0178) Administered by Intramuscular Route Versus Standard-Dose Quadrivalent Influenza Vaccine by Subcutaneous Route in Subjects 60 Years of Age and Older in Japan
Brief Title: Study to Assess the Immune Response and the Safety Profile of a High-Dose Quadrivalent Influenza Vaccine (QIV-HD) Compared to a Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD) in Japanese Adults 60 Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15150; U1111-1225-1085 (Other: UTN); QHD00010 (Other: Sanofi Pasteur)
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunization; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Participants randomized in each group were stratified by site and age (60 to 64, 65 to 74, and 75 years of age and older).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind: the participant and the Investigator remain unaware of the treatment assignments throughout the study. An unblinded qualified trial staff member will administer the appropriate vaccine but will not be involved in the immunogenicity and safety evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: QIV-HD (Experimental): Participants received a single injection of 0.7 milliliters (mL) high dose quadrivalent influenza vaccine (QIV-HD), intramuscularly (IM) at Day 0.
  Interventions: Biological: High-Dose Quadrivalent Influenza Vaccine, (Zonal Purified, Split Virus) 2020-2021 Strains (QIV-HD)
- Group 2: QIV-SD (Active Comparator): Participants received a single injection of 0.5 mL standard-dose quadrivalent influenza vaccine (QIV-SD), subcutaneously (SC) at Day 0.
  Interventions: Biological: Local Standard-Dose Inactivated Quadrivalent Influenza Vaccine, 2020-2021 Strains (QIV-SD)

INTERVENTIONS:
Biological: High-Dose Quadrivalent Influenza Vaccine, (Zonal Purified, Split Virus) 2020-2021 Strains (QIV-HD) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: IM
  Other Names: QIV-HD
  Arms: Group 1: QIV-HD
Biological: Local Standard-Dose Inactivated Quadrivalent Influenza Vaccine, 2020-2021 Strains (QIV-SD) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: SC
  Other Names: QIV-SD
  Arms: Group 2: QIV-SD

SUMMARY:
Primary Objective:

To demonstrate that QIV-HD induced an immune response (as assessed by hemagglutination inhibition [HAI] geometric mean titers [GMTs] and seroconversion rates) that was superior to responses induced by QIV-SD for the 4 virus strains at 28 days post-vaccination in all participants.

Secondary Objective:

* To describe the immune response induced by QIV-HD and QIV-SD by HAI measurement method in all participants.
* To describe the safety profile of all participants in each study group.

DETAILED DESCRIPTION:
Study duration per participant was approximately 28 days including: 1 day of screening and vaccination, a safety follow-up telephone call and an end of study visit approximately at Day 8 and 28 after vaccination, respectively.

ELIGIBILITY:
Inclusion criteria :

* Aged greater than or equal to (>=) 60 years on the day of inclusion.
* Able to attend all scheduled visits and complied with all study procedures.

Exclusion criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccination with live vaccines within the past 27 days preceding the study vaccination or any vaccination with inactivated vaccines within the past 6 days preceding the study vaccination, or planned receipt of any vaccine prior to Visit 02.
* Previous vaccination against influenza (in the preceding 6 months) with either the study vaccine or another vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the study or to a vaccine containing any of the same substances.
* Thrombocytopenia or bleeding disorder, contraindicating IM vaccination based on Investigator's judgment.
* Alcohol or substance abuse that, in the opinion of the Investigator might interfere with the study conduct or completion.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e.,parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Personal or family history of Guillain-Barré syndrome.
* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy and participants who have a history of neoplastic disease and have been disease free for >=5 years).
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >=37.5 degree Celsius). A prospective participant was not be included in the study until the condition had resolved or the febrile event had subsided.
* History of convulsions.
* Any condition that in the opinion of the Investigator could interfere with the evaluation of the vaccine.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2100 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- Japan (10):
  - Investigational Site Number 3920005, Fukuoka
  - Investigational Site Number 3920004, Koganeishi
  - Investigational Site Number 3920006, Kumamoto
  - Investigational Site Number 3920001, Osaka
  - Investigational Site Number 3920003, Shinjuku-Ku
  - Investigational Site Number 3920008, Shinjuku-Ku
  - Investigational Site Number 3920009, Shinjuku-Ku
  - Investigational Site Number 3920002, Suita-Shi
  - Investigational Site Number 3920007, Toshima-Ku
  - Investigational Site Number 3920010, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Sanchez L, Nakama T, Nagai H, Matsuoka O, Inoue S, Inoue T, Shrestha A, Pandey A, Chang LJ, De Bruijn I; QHD00010 Study Group. Superior immunogenicity of high-dose quadrivalent inactivated influenza vaccine versus Standard-Dose vaccine in Japanese Adults >/= 60 years of age: Results from a phase III, randomized clinical trial. Vaccine. 2023 Apr 6;41(15):2553-2561. doi: 10.1016/j.vaccine.2023.02.071. Epub 2023 Mar 10. PMID 36906404
- See also: EFC15150 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25229&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 active centers in Japan.
Pre-assignment Details: A total of 2100 participants were enrolled and randomized between 21 October 2020 to 14 January 2021.
Groups:
- QIV-HD: Participants received a single injection of 0.7 milliliters (mL) high dose quadrivalent influenza vaccine (QIV-HD), intramuscularly (IM) at Day 0.
- QIV-SD: Participants received a single injection of 0.5 mL standard-dose quadrivalent influenza vaccine (QIV-SD), subcutaneously (SC) at Day 0.
Period: Overall Study
Arm/Group | QIV-HD | QIV-SD
Started | 1049 | 1051
Completed | 1048 | 1047
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Arm/Group | QIV-HD | QIV-SD | Total Title
Number analyzed (Participants) | 1049 | 1051 | 2100
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (4.89) | 68.4 (4.96) | 68.3 (4.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 486 | 504 | 990
  Male | 563 | 547 | 1110
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1049 | 1051 | 2100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies at Day 28
Description: GMTs of anti-influenza antibodies were measured using hemagglutination inhibition (HAI) assay for 4 influenza virus strains: A/H1N1, A/H3N2-like, B/Victoria-like, and B/Yamagata. Titers were expressed in terms of 1/dilution.
Time Frame: Day 28 (post-vaccination)
Population: Analysis was performed on full analysis set (FAS) population which included all randomized participants who received at least one dose of the study vaccine and had a post-vaccination blood sample HAI result for at least one strain. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1048 | 1047
titers
  A/H1N1 | 309.0 [282.1 to 338.4] | 110.0 [100.0 to 121.1]
  A/H3N2-like: number analyzed (Participants) | 1048 | 1046
  A/H3N2-like | 540.0 [504.4 to 578.0] | 239.9 [222.0 to 259.1]
  B/Victoria-like | 354.8 [333.0 to 378.0] | 139.2 [129.4 to 149.8]
  B/Yamagata | 795.8 [750.3 to 844.1] | 254.7 [237.7 to 273.0]
Statistical Analysis 1: Comparison: QIV-HD vs QIV-SD; A/H1N1; Test type: Superiority — Superiority of GMTs was concluded if the lower limit of the 2-sided 95% Confidence Interval (CI) for the ratio of GMTs was greater than (>) 1 between groups for each of the comparisons; GMT ratio = 2.81, 95% CI 2-sided [2.46 to 3.20] — The 2-sided 95% CI was based on the student t-distribution of logarithmic transformation of the individual titers. Antilog transformations were applied to the results
Statistical Analysis 2: Comparison: QIV-HD vs QIV-SD; A/H3N2-like; Test type: Superiority — Superiority of GMTs was concluded if the lower limit of the 2-sided 95%CI for the ratio of GMTs was >1 between groups for each of the comparisons; GMT ratio = 2.25, 95% CI 2-sided [2.03 to 2.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: QIV-HD vs QIV-SD; B/Victoria-like; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 2.55, 95% CI 2-sided [2.31 to 2.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: QIV-HD vs QIV-SD; B/Yamagata; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 3.12, 95% CI 2-sided [2.85 to 3.42] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Participants Achieving Seroconversion Against Influenza Virus Antigens: Superiority Analysis
Description: Anti-influenza antibodies were measured by HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2-like, B/Victoria-like, and B/Yamagata. Seroconversion was defined as either a pre-vaccination HAI titer less than (<) 10 (1/dilution) and a post-vaccination titer >=40 (1/dilution) or a pre-vaccination titer >=10 (1/dilution) and a >= four-fold increase in post-vaccination titer at Day 28.
Time Frame: Day 28 (post-vaccination)
Population: Analysis was performed on FAS population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1048 | 1047
percentage of participants
  A/H1N1: number analyzed (Participants) | 1045 | 1045
  A/H1N1 | 77.6 [75.0 to 80.1] | 47.9 [44.9 to 51.0]
  A/H3N2-like: number analyzed (Participants) | 1047 | 1045
  A/H3N2-like | 75.4 [72.6 to 77.9] | 47.3 [44.2 to 50.4]
  B/Victoria-like: number analyzed (Participants) | 1046 | 1045
  B/Victoria-like | 79.2 [76.6 to 81.6] | 47.8 [44.7 to 50.8]
  B/Yamagata: number analyzed (Participants) | 1045 | 1045
  B/Yamagata | 74.4 [71.7 to 77.1] | 39.0 [36.1 to 42.1]
Statistical Analysis 1: Comparison: QIV-HD vs QIV-SD; A/H1N1; Test type: Superiority — Superiority on seroconversions was concluded if the lower limit of the 2-sided 95% CI of the difference in percentage between groups was > 0% for each of the comparisons; Difference in percentage = 29.7, 95% CI 2-sided [25.7 to 33.5] — The 2-sided 95% CI for the difference was based on the Wilson score method without continuity correction
Statistical Analysis 2: Comparison: QIV-HD vs QIV-SD; A/H3N2-like; Test type: Superiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = 28.1, 95% CI 2-sided [24.0 to 32.0] — The 2-sided 95% CI for the difference was based on the Wilson score method without continuity correction
Statistical Analysis 3: Comparison: QIV-HD vs QIV-SD; B/Victoria-like; Test type: Superiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = 31.4, 95% CI 2-sided [27.4 to 35.2] — The 2-sided 95% CI for the difference was based on the Wilson score method without continuity correction
Statistical Analysis 4: Comparison: QIV-HD vs QIV-SD; B/Yamagata; Test type: Superiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = 35.4, 95% CI 2-sided [31.4 to 39.3] — The 2-sided 95% CI for the difference was based on the Wilson score method without continuity correction

3. Secondary Outcome: GMTs of Influenza Vaccine Antibodies at Day 0 and Day 28
Description: GMTs of anti-influenza antibodies were measured using HAI assay for 6 influenza virus strains: A/H1N1, A/H3N2, A/H3N2-like, B/Victoria, B/Victoria-like, and B/Yamagata. Titers were expressed in terms of 1/dilution.
Time Frame: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1048 | 1047
titers
  A/H1N1: Day 0: number analyzed (Participants) | 1045 | 1045
  A/H1N1: Day 0 | 14.5 [13.5 to 15.5] | 14.9 [13.9 to 16.1]
  A/H1N1: Day 28 | 309.0 [282.1 to 338.4] | 110.0 [100.0 to 121.1]
  A/H3N2: Day 0: number analyzed (Participants) | 1047 | 1045
  A/H3N2: Day 0 | 54.9 [50.3 to 59.9] | 54.6 [50.0 to 59.7]
  A/H3N2: Day 28 | 721.4 [676.6 to 769.2] | 319.9 [297.1 to 344.5]
  A/H3N2-like: Day 0: number analyzed (Participants) | 1047 | 1045
  A/H3N2-like: Day 0 | 40.8 [37.5 to 44.4] | 41.0 [37.6 to 44.7]
  A/H3N2-like: Day 28: number analyzed (Participants) | 1048 | 1046
  A/H3N2-like: Day 28 | 540.0 [504.4 to 578.0] | 239.9 [222.0 to 259.1]
  B/Victoria: Day 0: number analyzed (Participants) | 1046 | 1045
  B/Victoria: Day 0 | 26.3 [24.4 to 28.3] | 24.7 [23.0 to 26.5]
  B/Victoria: Day 28 | 447.3 [420.8 to 475.5] | 152.0 [141.4 to 163.4]
  B/Victoria-like: Day 0: number analyzed (Participants) | 1046 | 1045
  B/Victoria-like: Day 0 | 23.7 [22.1 to 25.5] | 22.3 [20.9 to 23.9]
  B/Victoria-like: Day 28 | 354.8 [333.0 to 378.0] | 139.2 [129.4 to 149.8]
  B/Yamagata: Day 0: number analyzed (Participants) | 1045 | 1045
  B/Yamagata: Day 0 | 70.4 [64.4 to 77.1] | 60.4 [55.3 to 66.0]
  B/Yamagata: Day 28 | 795.8 [750.3 to 844.1] | 254.7 [237.7 to 273.0]

4. Secondary Outcome: Geometric Mean Titers Ratio (GMTR) of Influenza Vaccine Antibodies
Description: GMTs of anti-influenza antibodies were measured using HAI assay for 6 influenza virus strains: A/H1N1, A/H3N2, A/H3N2-like, B/Victoria, B/Victoria-like, and B/Yamagata. GMTRs were calculated as the ratio of GMTs post-vaccination (on Day 28) and pre-vaccination (on Day 0).
Time Frame: Day 0 (pre-vaccination), Day 28 (post-vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1048 | 1047
ratio
  A/H1N1: number analyzed (Participants) | 1045 | 1045
  A/H1N1 | 21.33 [19.57 to 23.25] | 7.33 [6.71 to 8.01]
  A/H3N2: number analyzed (Participants) | 1047 | 1045
  A/H3N2 | 13.14 [12.05 to 14.32] | 5.86 [5.34 to 6.42]
  A/H3N2-like: number analyzed (Participants) | 1047 | 1045
  A/H3N2-like | 13.23 [12.13 to 14.43] | 5.85 [5.33 to 6.42]
  B/Victoria: number analyzed (Participants) | 1046 | 1045
  B/Victoria | 17.06 [15.78 to 18.44] | 6.17 [5.66 to 6.72]
  B/Victoria-like: number analyzed (Participants) | 1046 | 1045
  B/Victoria-like | 14.97 [13.88 to 16.14] | 6.27 [5.76 to 6.82]
  B/Yamagata: number analyzed (Participants) | 1045 | 1045
  B/Yamagata | 11.29 [10.39 to 12.27] | 4.21 [3.88 to 4.57]

5. Secondary Outcome: Percentage of Participants Achieving Seroconversion Against Influenza Virus Antigens
Description: Anti-influenza antibodies were measured by HAI assay for 6 influenza virus strains: A/H1N1, A/H3N2, A/H3N2-like, B/Victoria, B/Victoria-like, and B/Yamagata. Seroconversion was defined as either a pre-vaccination HAI titer <10 (1/dilution) and a post-vaccination titer >=40 (1/dilution) or a pre-vaccination titer >=10 (1/dilution) and a >= four-fold increase in post-vaccination titer at Day 28.
Time Frame: Day 28 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1048 | 1047
percentage of participants
  A/H1N1: number analyzed (Participants) | 1045 | 1045
  A/H1N1 | 77.6 [75.0 to 80.1] | 47.9 [44.9 to 51.0]
  A/H3N2: number analyzed (Participants) | 1047 | 1045
  A/H3N2 | 76.4 [73.7 to 79.0] | 48.2 [45.2 to 51.3]
  A/H3N2-like: number analyzed (Participants) | 1047 | 1045
  A/H3N2-like | 75.4 [72.6 to 77.9] | 47.3 [44.2 to 50.4]
  B/Victoria: number analyzed (Participants) | 1046 | 1045
  B/Victoria | 82.1 [79.7 to 84.4] | 47.4 [44.3 to 50.4]
  B/Victoria-like: number analyzed (Participants) | 1046 | 1045
  B/Victoria-like | 79.2 [76.6 to 81.6] | 47.8 [44.7 to 50.8]
  B/Yamagata: number analyzed (Participants) | 1045 | 1045
  B/Yamagata | 74.4 [71.7 to 77.1] | 39.0 [36.1 to 42.1]

6. Secondary Outcome: Percentage of Participants With HAI Titers >=40 (1/Dilution) Against Influenza Antigens
Description: Anti-influenza antibodies were measured using HAI assay method for 6 influenza virus strains: A/H1N1, A/H3N2, A/H3N2-like, B/Victoria, B/Victoria-like, and B/Yamagata. Percentage of participants with HAI titers >=40 (1/dilution) is reported in the outcome measure.
Time Frame: Day 0 (pre-vaccination), Day 28 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1048 | 1047
percentage of participants
  A/H1N1: Day 0: number analyzed (Participants) | 1045 | 1045
  A/H1N1: Day 0 | 16.1 [13.9 to 18.4] | 18.2 [15.9 to 20.7]
  A/H1N1: Day 28 | 85.1 [82.8 to 87.2] | 67.6 [64.7 to 70.5]
  A/H3N2: Day 0: number analyzed (Participants) | 1047 | 1045
  A/H3N2: Day 0 | 52.3 [49.3 to 55.4] | 51.7 [48.6 to 54.7]
  A/H3N2: Day 28 | 98.9 [98.0 to 99.4] | 93.4 [91.7 to 94.8]
  A/H3N2-like: Day 0: number analyzed (Participants) | 1047 | 1045
  A/H3N2-like: Day 0 | 43.9 [40.9 to 47.0] | 43.7 [40.7 to 46.8]
  A/H3N2-like: Day 28: number analyzed (Participants) | 1048 | 1046
  A/H3N2-like: Day 28 | 96.8 [95.5 to 97.7] | 88.4 [86.3 to 90.3]
  B/Victoria: Day 0: number analyzed (Participants) | 1046 | 1045
  B/Victoria: Day 0 | 29.7 [27.0 to 32.6] | 27.8 [25.1 to 30.7]
  B/Victoria: Day 28 | 97.9 [96.8 to 98.7] | 81.4 [78.9 to 83.7]
  B/Victoria-like: Day 0: number analyzed (Participants) | 1046 | 1045
  B/Victoria-like: Day 0 | 25.1 [22.5 to 27.9] | 24.1 [21.5 to 26.8]
  B/Victoria-like: Day 28 | 96.8 [95.5 to 97.7] | 79.8 [77.2 to 82.1]
  B/Yamagata: Day 0: number analyzed (Participants) | 1045 | 1045
  B/Yamagata: Day 0 | 60.6 [57.5 to 63.6] | 56.9 [53.9 to 60.0]
  B/Yamagata: Day 28 | 98.9 [98.0 to 99.4] | 92.3 [90.5 to 93.8]

7. Secondary Outcome: Number of Participants Reporting Immediate Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or in a clinical investigation participant administered a medicinal product and which did not necessarily have a casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. All participants were observed for 30 minutes after vaccination, and any unsolicited AEs that occurred during that time were recorded as immediate unsolicited AEs in the CRB.
Time Frame: Within 30 minutes post-vaccination
Population: Analysis was performed on safety analysis set (SafAS) population which included participants who had received the study vaccine and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1049 | 1051
Participants | 0 | 1

8. Secondary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRB and considered as related to the product administered. Solicited injection site reactions included injection site pain, injection site erythema, injection site swelling, injection site induration, and injection site bruising. Solicited systemic reactions included fever, headache, malaise, myalgia and shivering.
Time Frame: Within 7 days post-vaccination
Population: Analysis was performed on the SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1049 | 1051
Participants
  Injection site pain | 503 | 334
  Injection site erythema | 86 | 328
  Injection site swelling | 82 | 185
  Injection site induration | 52 | 107
  Injection site bruising | 5 | 11
  Fever | 8 | 1
  Headache | 105 | 75
  Malaise | 102 | 59
  Myalgia | 197 | 130
  Shivering | 51 | 25

9. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or in a clinical investigation participant administered a medicinal product and which did not necessarily have a casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination.
Time Frame: Within 28 days post-vaccination
Population: Analysis was performed on SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1049 | 1051
Participants | 71 | 85

10. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: A SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event.
Time Frame: From Day 0 up to Day 28 post-vaccination
Population: Analysis was performed on the SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | QIV-HD | QIV-SD
Number analyzed (Participants) | 1049 | 1051
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: Unsolicited AEs were collected from Day 0 (post-vaccination) up to 28 days post-vaccination. Solicited reaction data were collected up to Day 7 post-vaccination. SAE data were collected from Day 0 up to Day 28 post-vaccination.
Description: Analysis was performed on the safety analysis set. A solicited reaction was an adverse reaction that was prelisted (i.e., solicited) in the CRB and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the CRB in terms of diagnosis and/or onset window post-vaccination.
Arm/Group | QIV-HD | QIV-SD
All-Cause Mortality (participants affected / at risk) | 0/1049 | 0/1051
Serious Adverse Events (participants affected / at risk) | 2/1049 | 5/1051
Other Adverse Events (participants affected / at risk) | 614/1049 | 569/1051
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QIV-HD (N=1049) | QIV-SD (N=1051)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Still's Disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QIV-HD (N=1049) | QIV-SD (N=1051)
Injection Site Erythema (General disorders) | 86 (86) | 328 (328)
Injection Site Induration (General disorders) | 52 (52) | 107 (107)
Injection Site Pain (General disorders) | 503 (504) | 334 (334)
Injection Site Swelling (General disorders) | 82 (82) | 185 (185)
Malaise (General disorders) | 102 (103) | 59 (59)
Myalgia (Musculoskeletal and connective tissue disorders) | 197 (197) | 130 (130)
Headache (Nervous system disorders) | 107 (108) | 76 (76) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT04498832/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04498832/SAP_001.pdf